CLINICAL TRIAL: NCT05114278
Title: Effect of Intravenous Iron Supplementation on Celiac Disease Remission in Patients With Iron Deficiency and Intestinal Villous Atrophy: a Randomized Trial
Brief Title: Effect of Intravenous Iron Supplementation on Celiac Disease Remission (IRONCEL)
Acronym: IRONCEL
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P170915J; 2019-003125-21 (EudraCT Number); PHRCN-17-0647 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2021-09-09; First posted 2021-11-09 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Iron deficiency
MeSH Terms: conditions — Celiac Disease; Iron Deficiencies | interventions — ferric carboxymaltose; Iron

STUDY DESIGN:
Intervention Model Description: Phase IV, open, randomized, 2-arms parallel controlled trial with blinded assessment of end-point.
Who Masked: Outcomes Assessor
Masking Description: Upper endoscopy with duodenal biopsy will be performed at most one month before randomization, and one month after the last infusion (experimental group) and between the 12th and the 13h month after randomization (control group). Histological analysis (villous recovery, primary endpoint) will be centrally performed by an expert pathologist blind to the group of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Iron + IV Ferinject (Experimental): Experimental group will receive intravenous iron infusion (Ferinject©: 15 mg/kg in NaCl solution IV) at randomization, 2weeks after randomization, 4weeks after randomization, and then every month for a total of one year.
  Interventions: Drug: Ferinject; Drug: oral iron
- Oral Iron only (Active Comparator): Comparison group will not receive any intravenous treatment. Both experimental and comparison groups will receive an oral iron supplementation (100 mg/day).
  Interventions: Drug: oral iron

INTERVENTIONS:
Drug: Ferinject — Experimental group will receive intravenous iron infusion (Ferinject©: 15 mg/kg in NaCl solution IV) at randomization, 2weeks after randomization, 4weeks after randomization, and then every month for a total of one year. Comparison group will not receive any intravenous treatment. Both experimental and comparison groups will receive an oral iron supplementation (100 mg/day).
  Other Names: Experimental arm
  Arms: Oral Iron + IV Ferinject
Drug: oral iron — All patients will receive an oral iron supplementation (100mg/day).
  Other Names: Control arm

SUMMARY:
The study aims is to evaluate the efficacy of intravenous iron supplementation on celiac disease remission (total intestinal mucosal recovery). This randomized multicenter trial compare the administration of intravenous iron by infusion (Ferinject©: 15 mg/kg in NaCl solution in 30 min) and oral iron in combination; to patients receive only oral iron as standard care.

The first benefit with IV Iron supplementation is to correct iron deficiency more rapidly than oral iron alone because of trouble of absorption in case of intestinal villous atrophy.

DETAILED DESCRIPTION:
Celiac disease is an autoimmune-like disorder induced in genetically predisposed individuals by dietary proteins from wheat (gluten). Its frequency reaches 1% in Europe.

In celiac patients, gluten induces small intestinal villous atrophy and, as a consequence, malnutrition. Celiac disease treatment relies on a long-life strict gluten-free diet that allows clinical and histological recovery and prevents long-term complications (autoimmune diseases, osteoporosis and malignancies). Remission is attested by total villous recovery on duodenal biopsy performed after one year of gluten free diet. Yet, in adults, systematic follow-up of biopsies for several years after gluten free diet initiation has recently revealed persistent villous atrophy in more than 40 % of cases with an increased risk in older patients (up to 56%). Lack of mucosal healing has been associated with the risk of complications in celiac, notably a risk factor for fractures and lymphoma. It is therefore necessary to define strategies to obtain and accelerate full recovery. Iron deficiency is strongly associated with celiac disease and is generally viewed as a consequence of small intestinal lesions and a symptom of malnutrition. Our preliminary clinical retrospective study showed more frequent iron deficiency anemia in celiac patients with (20/70; 29%) than without (11/88; 12.5%) villous atrophy (p = 0.015; OR: 2.78). Our previous experimental study suggests that iron deficiency may sustain tissue damage and delay mucosal recovery in celiac disease. Indeed the transferrin receptor (CD71) is overexpressed in the gut epithelium in case of iron deficiency and can interact with secretory IgA1 present in large amounts in the intestinal lumen of CD patients. Crosslinking of CD71 by polymeric IgA1 can induce production of inflammatory cytokines. Our working hypothesis is therefore that iron deficiency maintains aberrant expression of CD71 at the gut epithelial surface that sustains intestinal inflammation and epithelial damage. Iron supplementation of celiac patients with villous atrophy and iron deficiency may accelerate mucosal healing, villous recovery and remission.

ELIGIBILITY:
Inclusion Criteria:

* Patients free of mental illness, able to sign consent and >18year
* Celiac disease confirmed by presence of serum celiac antibodies and villous atrophy on intestinal biopsy before starting gluten free diet (GFD)
* Intestinal villous atrophy on duodenal biopsy (performed within 1 month) showing villous atrophy
* Patient under GFD or starting GFD with strict compliance
* Hemoglobin level (Hb) <12g/dL & Hb>8g/dL
* Well tolerated anemia
* Iron deficiency defined by: serum iron level < 11 µmol/L, ferritinemia < 20µg/L and/or transferrin saturation index <0.2

Exclusion Criteria:

* Patient not able to sign, mental illness, pregnancy
* Complicated celiac disease: intestinal malignancies
* Severe anemia (Hb <8g/dL) and/or poorly tolerated anemia requiring systematic iron IV supplementation or blood transfusion
* Serious severe disease having short-term prognostic implication
* Contraindication to intravenous iron infusion: known drug allergy
* Pregnant or breastfeeding women
* Participation in another interventional trial
* Patients treated by steroids, immunosuppressors or chemotherapy drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Total villous recovery | 12 months
  The primary endpoint is the proportion of patients with total villous recovery (total remission) on the last duodenal biopsies. 6 formalin and 2 frozen duodenal biopsies will be performed. Intestinal mucosal assessment will be performed by a centralized histological analysis according to the Marsh classification. Readers will be blind to the treatment received.

SECONDARY OUTCOMES:
Atrophic gastritis | 12 months
  Proportion of patients with atrophic gastritis at V0 and at V14 biopsies (2 in the antrum, 1 in the angulus and 2 in the fundus)
Partial recovery of intestinal villous atrophy | 12 months
  Proportion of patients with partial recovery of intestinal villous atrophy on the last control duodenal biopsies according to Marsh classification (centralized histological analysis). Six formalin and two frozen duodenal biopsies will be performed.
Iron deficiency | 12 months
  Proportion of patients correcting iron deficiency. Iron parameters (serum iron level (µmol/L), ferritinemia (µg/L), transferrin saturation index) will be assessed at visit V1, V3, V6, V10, V14; correction of iron deficiency is defined by serum iron level > 20 µg/L and transferrin saturation index ≥0.20.
Anaemia | 12 months
  Proportion of patients correcting anaemia during the 12 months participation. Hemoglobin (Hb) level (g/d) will be measured at visit V1, V3, V6, V10, V14. Correction of anaemia is defined by Hb≥12g/L in woman and Hb≥13g/dL in man.
Intraepithelial lymphocytes | 12 months
  Evolution of the count of intraepithelial lymphocytes assessed on initial and last control biopsy.
CD71 on epithelial cells | 12 months
  Evolution of the expression of CD71 on epithelial cells studied on initial and last control biopsy
Body Mass Index | 12 months
  Evolution of the patient's BMI during his participation at the study.
Serum folate level | 12 months
  Serum folate level (µg/L) measured at visit V1, V3, V6, V10, V14.
Vitamin B12 level | 12 months
  Level of vitamin B12 (pmol/L) measured at visit V1, V3, V6, V10, V14.
Calcemia level | 12 months
  Level of calcemia (mmol/L) measured at visit V1, V3, V6, V10, V14.
Albuminemia level | 12 months
  Level of albuminemia (g/L) measured at visit V1, V3, V6, V10, V14.
Corrected calcemia level | 12 months
  Level of corrected calcemia (mmol/L) measured at visit V1, V3, V6, V10, V14.
25(OH)D3 vitamin level | 12 months
  Level of 25(OH)D3 vitamin measured at visit V1, V3, V6, V10, V14.
Liver enzymes | 12 months
  Evolution of serum levels of liver enzymes (AST, ALT, AP, gGT, Total Bilirubin), glycemia, T4, TSH measured at visit V1, V3, V6, V10, V14.
Gluten free diet | 12 months
  Observance of gluten free diet will be assessed by (i) dietitian assessment of gluten free consumption (g/day and proportion of patients in high (0 g/day), medium (0-50 mg/day), low (>50 mg/day) observance), (ii) measurement of serum celiac antibodies (anti-tTG IgA and anti-deamidated gliadin IgG) and (iii) proportion of patients having gluten immunogenic peptides excretion detected in urine at visit V1, V3, V6,V10, V14.
Patient quality of life | 12 months
  French Celiac disease questionnaire assessed at V1 and V14 about the evolution of the quality of life for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia MALAMUT, MD, PhD, Principal Investigator — Cochin, AP-HP, Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and PI team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).